CLINICAL TRIAL: NCT03809325
Title: Cross-sectional Survey to Collect Treatment Experience Feedback From Patients, Physicians, Nurses and Carers After Switching to Paliperidone Palmitate 3-monthly
Brief Title: A Survey to Collect Treatment Experience Feedback From Patients, Physicians, Nurses and Carers After Switching to Paliperidone Palmitate 3-monthly
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108568; R092670SCH4066 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Schizophrenia: No intervention will be administered as a part of this study. Participants diagnosed with schizophrenia, who have been treated with 4 to 6 injections of paliperidone palmitate 3-month formulation (PP3M), together with the corresponding physician, and the corresponding nurse and carer where applicable for each participant will be enrolled in this survey. The data source for this study will be the online questionnaire used for each participant, physician, and the corresponding nurse and carer where applicable.
  Interventions: Drug: Paliperidone Palmitate 3-Month Formulation (PP3M)

INTERVENTIONS:
Drug: Paliperidone Palmitate 3-Month Formulation (PP3M) — No intervention will be administered as a part of this study. Participants who have been treated with PP3M in clinical practice will be enrolled.
  Other Names: Trevicta

SUMMARY:
The purpose of this study is to explore the experience with paliperidone palmitate 3-month formulation (PP3M) treatment of participants and their corresponding physicians, nurses and carers, to understand the impact of less frequent injections from their perspective.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenia (according to International Classification of Diseases [ICD]-10)
* Be currently receiving PP3M and have previously received 4 to 6 injections of PP3M
* Have the required language skills to participate in the online questionnaire, in the opinion of the physician
* Be able and willing to provide their informed consent for study participation

Exclusion Criteria:

* Has received involuntary treatment with PP3M
* Was switched to PP3M treatment within a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with schizophrenia who are currently receiving paliperidone palmitate 3-month formulation (PP3M) and have previously received 4 to 6 injections of PP3M treatment will be enrolled. Feedback will be collected using an online questionnaire-based tool at a single data collection time point.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Participant's Experience with PP3M Treatment | 1 day
  Participant's experience with paliperidone palmitate 3-month formulation (PP3M) treatment will be evaluated qualitatively through an online questionnaire. Each questionnaire will include a total of approximately 30 to 35 multiple choice questions related to following categories: Impact on relationship/ interaction between medical team and carer/ patient, Involvement in treatment decision, Reasons for PP3M, Impact of treatment on patient, Impact of treatment on carer and General experience with PP3M.

SECONDARY OUTCOMES:
Responses to the Questionnaires | 1 day
  The response to the questionnaires of the corresponding physician, and the corresponding nurse and carer where applicable, for each participant will be collected for the following categories: Impact on relationship/ interaction between medical team and carer/ patient, Involvement in treatment decision, Reasons for PP3M, Impact of treatment on patient, Impact of treatment on carer and General experience with PP3M.
Clinical Global Impression-Severity (CGI-S) Score | 1 day
  The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. The CGI-S permits a global evaluation of the participant's condition at a given time.
Positive and Negative Syndrome Scale (PANSS) - Lack of Judgement and Insight's Score (G12 Item) | 1 day
  The PANSS is a validated scale specific for the measurement of the symptoms of schizophrenia. The neuropsychiatric symptoms of schizophrenia are assessed across 3 subscales comprising a total of 30 items; the positive [P] and negative [N] subscales each includes 7 items, while the general psychopathology [G] subscale includes 16 items. Lack of judgment and insight's score is 12th item of the general psychopathology subscale (G12 item) of PANSS with score ranges from 1 to 7. Higher scores indicate worsening.
European Quality of Life (EuroQol) 5-Dimension 5-Level (EQ 5D-5L) Questionnaire General Health Status Score | 1 day
  EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The responses to the 5 dimensions are used to compute a single utility score ranging from zero (worst health state) to 1 (better health state) representing the general health status of the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (41):
- Chu Brugmann, Brussels, Belgium
- France (11):
  - Centre Médico Psychologique De Courbevoie, Asnières-sur-Seine
  - Centre Medico Psychologique, Cagnes-sur-Mer
  - Cabinet medical, Dax
  - Centre Hospitalier Esquirol, Limoges
  - CH de Jury, Metz
  - CH Montauban, Montauban
  - Hopital la Colombiere, Montpellier
  - Centre Medico Psychologique Le Rembrandt, Nice
  - Centre Hospitalier de Novillars, Novillars
  - Centre Hospitalier Guillaume Regnier, Rennes
  - Hopital Sainte Musse, Toulon
- Germany (3):
  - Vivantes Klinikum Am Urban, Berlin
  - NPZR - Neuropsychatrisches Zentrum Riem, München
  - Kbo-Inn-Salzach-Klinikum GmbH, Wasserburg A. Inn
- Hungary (4):
  - Toldy Ferenc Kórház-Rendelőintézet, Cegléd
  - Kemenesaljai Egyesített Kórház-Szakorvosi Rendelointézet, Celldömölk
  - Sántha Kálmán Szakkórház, Nagykálló
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Italy (6):
  - Azienda Sanitaria Alto Adige, Bolzano
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia Presidio Spedali Civili, Brescia
  - CSM Frosinone, Frosinone
  - Casa di Cura Villa Von Siebenthal, Genzano di Roma
  - Centro Igiene Mentale ASL Salerno, Oliveto Citra
  - SPDC Asltaranto, Statte
- Spain (13):
  - Hosp. Abente E Lago, A Coruña
  - Csm Miraflores, Alcobendas
  - Csm Arganda Del Rey, Arganda
  - Usmc Carmona, Carmona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Usmc Mairena Del Aljarafe, Mairena del Aljarafe
  - Centre Hosp. de Manresa, Manresa
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. de Torrevieja, Torrevieja
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Csm Rondilla, Valladolid
  - Hosp. Psiquiatrico Alava, Vitoria-Gasteiz
  - Hosp. Univ. Miguel Servet, Zaragoza
- United Kingdom (3):
  - Birmingham & Solihull MH NHS FT, Birmingham
  - Leicester Partnership NHS Trust, Leicester
  - West London Mental Health Trust, London

IPD SHARING:
Plan to Share IPD: No